CLINICAL TRIAL: NCT07053423
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Dupilumab on Airway Inflammation Through Assessments of Mucus Plugging and Other Lung Imaging Parameters in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: A Study to Investigate Airway Inflammation With Dupilumab Subcutaneously in Participants Aged ≥40 to ≤85 Years With Chronic Obstructive Pulmonary Disease.
Acronym: AEOLUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS18583; 2025-521268-37 (Registry Identifier: CTIS); U1111-1314-5262 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form:Solution for injection-Route of administration:SC injection
  Other Names: SAR231893; Dupixent
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form:Solution for injection-Route of administration:SC injection
  Arms: Placebo

SUMMARY:
LPS18583 is a multinational, randomized, double-blind, placebo-controlled, parallel-group, Phase 4 study with 2 treatment groups. The purpose of this study is to assess the effect of dupilumab compared with placebo on airway inflammation, resistance, and remodeling including mucus plugging and its association with improvement on lung function, exacerbations, and quality of life improvement in participants aged 40 years of age up to 85 years of age (inclusive).

Study details include:

The study duration will be up to 40 weeks. The treatment duration will be up to 24 weeks. The number of visits will be 9.

ELIGIBILITY:
Inclusion Criteria:

Participants with a physician diagnosis of Chronic Obstructive Pulmonary Disease (COPD) who meet the following criteria at screening:

* Current or former smokers with a smoking history of ≥10 pack-years
* Moderate-to-severe COPD (post-BD FEV1/FVC ratio <0.70 and post-BD FEV1 % predicted >30% and ≤70%)
* Medical Research Council Dyspnea Scale grade ≥2 or COPD assessment test (CAT) score ≥10
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) category E , Frequent or severe exacerbations
* Background triple therapy (ICS + LABA + LAMA) for 3 months before randomization with a stable dose of medication for ≥1 month before Visit 1; dual therapy (LABA + LAMA) allowed if ICS is contraindicated
* Evidence of Type 2 inflammation: Participants with blood eosinophils ≥300 cells/μL at screening or with blood eosinophils ≥150 cells/μL at Visit 1 (screening) and with a history of blood eosinophils ≥300 cells/μL within the past year during stable state (non-exacerbation).
* Mucus score cutoff of ≥3

Exclusion Criteria:

* A current diagnosis of asthma according to the Global Initiative for Asthma diagnostic (GINA) guidelines, or documented history of asthma
* Significant pulmonary disease other than COPD (eg, lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome) or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts
* Treatment with oxygen >4.0 L/min for ≥8 hours/day Respiratory tract infection within 4 weeks before screening, or during the screening period
* Diagnosis of α-1 anti-trypsin deficiency
* Any biologic therapy (including experimental treatments and dupilumab)
* Participants on treatment with mucolytics unless on stable therapy for >6 months

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2028-12-23 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 24 in global lung mucus score (UCSF mucus scoring) | Baseline to Week 24
  The score is calculated by counting the number of bronchopulmonary segments which on CT scans contain at least one mucus plugs. The score ranges from 0 up to a maximum score of 18 corresponding to the 18 bronchopulmonary segments present in most people. In this system, a mucus plug is defined as a complete occlusion of the airway imaged at Total Lung Capacity (TLC). Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Change from baseline to Week 24 in mucus volume for global lung by High-resolution Computed Tomography (HRCT) | Baseline to Week 24
Change from baseline to Week 24 in trimmed distal airway wall thickness at TLC by HRCT | Baseline to Week 24
Change from baseline to Week 24 in airway resistance from R5 to R20 measured by Forced Oscillation Technique (FOT) | Baseline to Week 24
Change from baseline to Week 24 in Reactance area (AX) measured by FOT | Baseline to Week 24
Incidence of Treatment-Emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI) including potentially clinically significant abnormalities | Baseline to Week 36

CONTACTS AND LOCATIONS:
Locations (46):
- United States (4):
  - Finlay Medical Research- Site Number : 8400010, Miami, Florida
  - American Health Research - Charlotte- Site Number : 8400013, Charlotte, North Carolina
  - Clinical Research Associates of Central PA- Site Number : 8400002, DuBois, Pennsylvania
  - REX Clinical Trials - Beaumont- Site Number : 8400011, Beaumont, Texas
- Argentina (2):
  - Investigational Site Number : 0320001, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320003, Buenos Aires
- Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760002, Porto Alegre, Rio Grande do Sul, Brazil
- Denmark (2):
  - Investigational Site Number : 2080003, Aalborg
  - Investigational Site Number : 2080002, Vejle
- France (7):
  - Investigational Site Number : 2500008, La Tronche
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500005, Lyon
  - Investigational Site Number : 2500006, Marseille
  - Investigational Site Number : 2500002, Montpellier
  - Investigational Site Number : 2500003, Pessac
  - Investigational Site Number : 2500004, Reims
- Hungary (3):
  - Investigational Site Number : 3480003, Debrecen
  - Investigational Site Number : 3480001, Hajdúnánás
  - Investigational Site Number : 3480002, Pécs
- Italy (2):
  - Investigational Site Number : 3800001, Cona, Ferrara
  - Investigational Site Number : 3800004, Siena
- Netherlands (3):
  - Investigational Site Number : 5280001, Groningen
  - Investigational Site Number : 5280003, Hoofddorp
  - Investigational Site Number : 5280006, Nijmegen
- Poland (3):
  - Investigational Site Number : 6160001, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160003, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160002, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- South Korea (5):
  - Investigational Site Number : 4100005, Anyang-si, Gyeonggi-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Santander, Cantabria
  - Investigational Site Number : 7240002, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240004, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240003, Madrid
- Sweden (2):
  - Investigational Site Number : 7520002, Gothenburg
  - Investigational Site Number : 7520003, Lund
- Taiwan (2):
  - Investigational Site Number : 1580001, Kaohsiung City
  - Investigational Site Number : 1580002, Taipei
- United Kingdom (5):
  - Investigational Site Number : 8260002, Dundee, Dundee City
  - Investigational Site Number : 8260006, Newcastle upon Tyne, England
  - Investigational Site Number : 8260003, Leicester, Leicestershire
  - Investigational Site Number : 8260001, Bradford
  - Investigational Site Number : 8260009, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS18583 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26743&tenant=MT_SNY_9011